CLINICAL TRIAL: NCT07187401
Title: A Randomized, Double-Blind, Placebo-Controlled, First-In-Human Study of the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ALN-CFB, an Investigational siRNA Therapeutic Against Complement Factor B, in Participants With Paroxysmal Nocturnal Hemoglobinuria and Persistent Anemia on Approved C5-Inhibitor Therapy
Brief Title: A First-in-Human Safety and Efficacy Study of ALN-CFB, a Small Interfering RNA (siRNA) Targeting Complement Factor B, in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria With Persistent Anemia on a C5 Inhibitor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-CFB-PNH-2468; 2024-519806-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH); Persistent Anemia
Keywords: C5 inhibitor; Complement Factor B (CFB) protein; Red Blood Cells
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single-Ascending Dose Escalation (Experimental)
  Interventions: Drug: ALN-CFB
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-CFB — Administered as defined in the protocol
  Arms: Single-Ascending Dose Escalation
Drug: Placebo — Administered as defined in the protocol
  Arms: Placebo

SUMMARY:
This study is researching an experimental drug called ALN-CFB. The study is focused on people with Paroxysmal Nocturnal Hemoglobinuria (PNH) who are currently taking a complement component C5 inhibitor ("C5-inhibitor") and continue to have anemia (low red blood cell count).

The aim of the study is to see how tolerable ALN-CFB is compared to placebo. A placebo looks like the study drug but does not contain any drug.

The study is looking at several other research questions, including:

* What side effects may happen from taking ALN-CFB
* How much ALN-CFB is in the blood at different times
* How much Complement Factor B (CFB) protein levels in the blood are affected by ALN-CFB

DETAILED DESCRIPTION:
The protocol will be amended to describe Part B of the study after Part A data have been analyzed.

ELIGIBILITY:
Key Inclusion Criteria:

1. Has been diagnosed with PNH confirmed by a history of high flow cytometry from prior testing
2. Treated with a stable dose of C5 inhibitor (eculizumab or approved eculizumab biosimilar, ravulizumab, or crovalimab) for at least 24 weeks prior to screening visit, as described in the protocol
3. Has hemoglobin ≤10.5 g/dL at screening visit 1, with evidence of anemia prior to this visit, as described in the protocol
4. Has peripheral blood reticulocyte count of ≥100 x 10^9/L at screening visit 1

Key Exclusion Criteria:

1. Has history of bone marrow transplantation or receipt of an organ transplant
2. Has history of meningococcal infection or similar recurrent infections by other encapsulated bacterial organisms
3. Has any active, ongoing infection or a recent infection requiring ongoing systemic treatment with antibiotics, antivirals, or antifungals within 2 weeks of screening or during the screening period
4. Has laboratory evidence of bone marrow failure, as described in the protocol
5. Have recent, unstable medical conditions, not related to PNH or PNH-related complications, as described in the protocol

NOTE: Other Protocol Defined Inclusion / Exclusion Criteria Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2029-11-29 (Estimated); Study Completion 2031-07-15 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment-Emergent Adverse Events (TEAEs) | Through 365 Days
Severity of TEAEs | Through 365 Days

SECONDARY OUTCOMES:
Concentrations of combined ALN-CFB and major metabolites in plasma | Through 365 Days
Concentrations of combined ALN-CFB and major metabolites in urine | Through 24 Hours following ALN-CFB administration
Absolute change from baseline in CFB concentration | Baseline, Through 365 Days
Percentage change from baseline in CFB concentration | Baseline, Through 365 Days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- Toronto General Hospital, Toronto, Ontario, Canada
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/